CLINICAL TRIAL: NCT06065774
Title: Comparative Evaluation of Laterally Closed Tunnel (LCT) Technique and Modified Coronally Advanced Tunnel (MCAT) Technique in the Treatment of Isolated Gingival Recession: Randomized Controlled Clinical Trial
Brief Title: Comparing Two Different Tunneling Technique for Gingival Recession Treatment Using Two Different Matertial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elbana, Assistant Lecturer,Oral Medicine, Periodontology, Diagnosis and Oral Radiology Department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A04060722
Record Dates: First submitted 2023-09-13; First posted 2023-10-04 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Gingival Recession, Localized
Keywords: gingival recession; laterally closed tunnel; modified coronally advanced tunnel; porcine derived collagen matrix; isolated gingival recession; tunneling technique
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: The patients will be assigned into four treatment groups Group I comprises of patient undergoing The Laterally Closed Tunnel Technique with SCTG , Group II comprises of patients undergoing The Laterally Closed Tunnel Technique with collagen matrix mucograft , Group III comprises of patients undergoing Modified Coronally Advanced Tunnel Technique with SCTG and Group IV comprises of patients undergoing Modified Coronally Advanced Tunnel Technique with collagen matrix mucograft
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The Laterally Closed Tunnel Technique with SCTG (Experimental): An aseptic field was required for all surgical procedures using povidine iodine. Local anesthesia using 4% articane with 1:100.000 epinephrine was applied.•
  * Then specially designed tunneling instruments [devmed] were used through the sulcular incision to create a pouch.
  * A microsurgical blade was used at the inner surface of the pouch till sufficient tissue release was achieved.
  * Tissue forceps was used to approximate the mesial and distal margin of the gingiva at the pouch margin.
  * After harvesting the graft, it was placed at the prepared pouch after root surface biomodification using EDTA gel 24% for 2 minutes and copious rinsing with saline solution.
  * SCTG was pulled using single or mattress sutures and the graft was fixed mesial and distal at the inner part of the pouch using resorbable suture material [Vicryl suture], then the graft was sutured around the neck of the CEJ by sling suture 6/0 polypropylene.
  Interventions: Procedure: The Laterally Closed Tunnel Technique with SCTG; Drug: The Laterally Closed Tunnel Technique with collagen matrix mucograft; Procedure: Modified Coronally Advanced Tunnel Technique with SCTG.; Drug: Modified Coronally Advanced Tunnel Technique with collagen matrix mucograft
- The Laterally Closed Tunnel Technique with collagen matrix mucograft (Experimental): An aseptic field was required for all surgical procedures using povidine iodine. Local anesthesia using 4% articane with 1:100.000 epinephrine was applied.•
  * Then specially designed tunneling instruments [devmed] were used through the sulcular incision to create a pouch.
  * A microsurgical blade was used at the inner surface of the pouch till sufficient tissue release was achieved.
  * Tissue forceps was used to approximate the mesial and distal margin of the gingiva at the pouch margin.
  * After harvesting the graft, it was placed at the prepared pouch after root surface biomodification using EDTA gel 24% for 2 minutes and copious rinsing with saline solution.
  * collagen matrix was pulled using single or mattress sutures and the graft was fixed mesial and distal at the inner part of the pouch using resorbable suture material [Vicryl suture], then the graft was sutured around the neck of the CEJ by sling suture 6/0 polypropylene.
  Interventions: Procedure: The Laterally Closed Tunnel Technique with SCTG; Drug: The Laterally Closed Tunnel Technique with collagen matrix mucograft; Procedure: Modified Coronally Advanced Tunnel Technique with SCTG.; Drug: Modified Coronally Advanced Tunnel Technique with collagen matrix mucograft
- Modified Coronally Advanced Tunnel Technique with SCTG. (Experimental): * Supraperiosteal incisions was extended to the mucosal level beyond the MGJ to allow sufficient tissue mobility and release.
  * The tunnel was extended in all directions around the recession defect to create a sufficient pouch for connective tissue graft stabilization.
  * The interdental papilla tunneling adjacent to the defect was a critical step for technique success.
  * Then perfect root planning was performed at the denuded root surface to remove the necrotic cementum at the accessible recession defect.
  * Subsequently palatal anesthesia was given to harvest palatal SCTG using deepitheliailized free gingival graft (FGG) technique.
  * SCTG was pulled using single or mattress sutures and the graft was fixed mesial and distal at the inner part of the pouch using resorbable suture material [Vicryl suture], then the graft was sutured around the neck of the CEJ by sling suture 6/0 polypropylene.
  Interventions: Procedure: The Laterally Closed Tunnel Technique with SCTG; Drug: The Laterally Closed Tunnel Technique with collagen matrix mucograft; Procedure: Modified Coronally Advanced Tunnel Technique with SCTG.; Drug: Modified Coronally Advanced Tunnel Technique with collagen matrix mucograft
- Modified Coronally Advanced Tunnel Technique with collagen matrix mucograft (Experimental): * Supraperiosteal incisions was extended to the mucosal level beyond the MGJ to allow sufficient tissue mobility and release.
  * The tunnel was extended in all directions around the recession defect to create a sufficient pouch for connective tissue graft stabilization.
  * The interdental papilla tunneling adjacent to the defect was a critical step for technique success.
  * Then perfect root planning was performed at the denuded root surface to remove the necrotic cementum at the accessible recession defect.
  * Subsequently palatal anesthesia was given to harvest palatal SCTG using deepitheliailized free gingival graft (FGG) technique.
  * collagen matrix was pulled using single or mattress sutures and the graft was fixed mesial and distal at the inner part of the pouch using resorbable suture material [Vicryl suture], then the graft was sutured around the neck of the CEJ by sling suture 6/0 polypropylene.
  Interventions: Procedure: The Laterally Closed Tunnel Technique with SCTG; Drug: The Laterally Closed Tunnel Technique with collagen matrix mucograft; Procedure: Modified Coronally Advanced Tunnel Technique with SCTG.; Drug: Modified Coronally Advanced Tunnel Technique with collagen matrix mucograft

INTERVENTIONS:
Procedure: The Laterally Closed Tunnel Technique with SCTG — Local anesthesia using 4% articane with 1:100.000 epinephrine was applied.•
  Then specially designed tunneling instruments [devmed] were used through the sulcular incision to create a pouch.
  A microsurgical blade was used at the inner surface of the pouch till sufficient tissue release was achieved.
  Tissue forceps was used to approximate the mesial and distal margin of the gingiva at the pouch margin.
  After harvesting the graft, it was placed at the prepared pouch after root surface biomodification using EDTA gel 24% for 2 minutes and copious rinsing with saline solution.
  SCTG was pulled using single or mattress sutures and the graft was fixed mesial and distal at the inner part of the pouch using resorbable suture material [Vicryl suture], then the graft was sutured around the neck of the CEJ by sling suture 6/0 polypropylene.
Drug: The Laterally Closed Tunnel Technique with collagen matrix mucograft — Local anesthesia using 4% articane with 1:100.000 epinephrine was applied.•
  Then specially designed tunneling instruments [devmed] were used through the sulcular incision to create a pouch.
  A microsurgical blade was used at the inner surface of the pouch till sufficient tissue release was achieved.
  Tissue forceps was used to approximate the mesial and distal margin of the gingiva at the pouch margin.
  After harvesting the graft, it was placed at the prepared pouch after root surface biomodification using EDTA gel 24% for 2 minutes and copious rinsing with saline solution.
  collagen matrix was pulled using single or mattress sutures and the graft was fixed mesial and distal at the inner part of the pouch using resorbable suture material [Vicryl suture], then the graft was sutured around the neck of the CEJ by sling suture 6/0 polypropylene.
Procedure: Modified Coronally Advanced Tunnel Technique with SCTG. — Supraperiosteal incisions was extended to the mucosal level beyond the MGJ to allow sufficient tissue mobility and release.
  The tunnel was extended in all directions around the recession defect to create a sufficient pouch for connective tissue graft stabilization.
  The interdental papilla tunneling adjacent to the defect was a critical step for technique success.
  Then perfect root planning was performed at the denuded root surface to remove the necrotic cementum at the accessible recession defect.
  Subsequently palatal anesthesia was given to harvest palatal SCTG using deepitheliailized free gingival graft (FGG) technique.
  SCTG was pulled using single or mattress sutures and the graft was fixed mesial and distal at the inner part of the pouch using resorbable suture material [Vicryl suture], then the graft was sutured around the neck of the CEJ by sling suture 6/0 polypropylene.
Drug: Modified Coronally Advanced Tunnel Technique with collagen matrix mucograft — Supraperiosteal incisions was extended to the mucosal level beyond the MGJ to allow sufficient tissue mobility and release.
  The tunnel was extended in all directions around the recession defect to create a sufficient pouch for connective tissue graft stabilization.
  The interdental papilla tunneling adjacent to the defect was a critical step for technique success.
  Then perfect root planning was performed at the denuded root surface to remove the necrotic cementum at the accessible recession defect.
  Subsequently palatal anesthesia was given to harvest palatal SCTG using deepitheliailized free gingival graft (FGG) technique.
  collagen matrix was pulled using single or mattress sutures and the graft was fixed mesial and distal at the inner part of the pouch using resorbable suture material [Vicryl suture], then the graft was sutured around the neck of the CEJ by sling suture 6/0 polypropylene.

SUMMARY:
The goal of this clinical trial is to compare two different tunneling surgical technique in treatment of gingival recession using two different materials.

Participants will be divided into four groups according to the treatments they'll be given.

DETAILED DESCRIPTION:
Comparative Evaluation of laterally Closed Tunnel (LCT) Technique and Modified Coronally Advanced Tunnel (MCAT) Technique in the treatment of isolated gingival recession: Randomized controlled clinical trial.

Proposal Submitted in Partial Fulfillment of the Requirements of Doctor of philosophy Degree in Oral Medicine and Periodontology BY Ahmed Mohamed El-Bana B.D.S, MSC (Mansoura University, 2014) Assistant lecturer at Oral Medicine, Periodontology, Oral Diagnosis and Radiology Department 2021

Gingiva represents one of the important defense barriers of the periodontium and any alteration of its conditions may result in detrimental effects on the stability of the periodontium. Gingival recession is a common mucogingival problem that is associated with apical migration of the gingival margin and exposure of the root surface.Various factors are associated with increased incidence of gingival recession such as plaque-induced inflammation, violation of the biological width of the gingiva, aggressive teeth brushing and high frenulum attachment.

Various surgical techniques were described for the treatment of gingival recession from which, the coronally advanced flap (CAF) is one of the most commonly used techniques for root coverage of miller class I, II. Many modifications of CAF have been used to get the best treatment outcomes. The CAF can be used alone or in combination with connective tissue graft [CTG], platelet rich fibrin , enamel matrix derivative or any other regenerative materials. Various systematic reviews have reported the efficacy of CAF as the gold standard protocol for gingival recession treatment especially if used with CTG.

Tension free healing is the main goal to get the ideal results of gingival recession correction, which was difficult to achieve with a coronal displacement of the tunnel. In addition, the vestibular depth distortion was related to the procedures due to tissue tension. Therefore new clinical approaches are warranted to be more predictable and to minimize the post-operative complications.

Recently, mucogingival surgeries have been extremely improved with many advanced surgical techniques to be minimally invasive and to get better outcomes for complex recession defects that are associated with soft and hard tissue defects.

The split-flap approach using tunneling technique is one of the approaches used to treat gingival recession. However, it was associated with a lot of difficulties and risks of flap perforation and graft necrosis during the healing process.To overcome such limitations, a modification of the techniques has been adopted as modified coronally advanced tunneling (MCAT) which can be either full orpartial thickness tunnel followed by displacing and moving the tissue in a coronal direction. The results of MCAT are predictable regarding the mean root coverage and recession depth reduction. The outcomes were also improved after using sub epithelium connective tissue graft (SCTG) under the tunnel to augment the keratinized attached gingiva and yield more stable outcomes on the long term basis.

Laterally closed tunnel technique (LCT) is a minimally invasive novel technique proposed by Sculean and Allen in 2018 for the management of isolated gingival recession. Tunneling instruments and micro blades are used to create a pouch that extends apically beyond the mucogingival junction and also extends mesially and distally away from the recession defect to dissect and separate the muscles and collagen fibers to allow lateral tissue displacement without tension or vestibular distortion.

Although the SCTG is the gold standard soft tissue graft and is associated with complete root coverage and ideal esthetics and maturation, it was associated with many tissue morbidities and healing complications. SCTG needs second surgical site which may be not accepted by many patients. Therefore many regenerative alterative tissue substitutes have been tested and investigated to be used in recession coverage surgeries instead of SCTG.

Mucoderm or porcine-derived collagen matrix has been used in many studies as an alternative to connective tissue graft CTG as a soft tissue grafting material for volume augmentation and gingival phenotype modification. Furthermore, it acts as a seeding scaffold on which cells can grow and differentiate into gingival fibroblasts. It has been investigated in many studies around teeth and dental implants with predictable outcomes.

Aim of the study

The objective of the current study is to compare two different surgical tunneling techniques: the laterally closed tunnel (LCT) and modified coronally advanced tunnel (MCAT) in the treatment of deep isolated gingival recession defects using subepithelial connective tissue graft (SCTG) and porcine derived collagen matrix (MUCODERM).

Material and methods

A total of 80 patients with isolated mandibular gingival recession defects will be selected from the outpatient clinic of the Department of Oral Medicine and Periodontology Department, Faculty of Dentistry, Mansoura University. The patients will be informed about the treatment protocol that they will receive and the steps that will be done. This includes the possible effects or risks, and other treatment options according to the rules of the ethical committee of the faculty of dentistry, Mansoura University. The subjects must understand this explanation in broad terms. The subjects must be legally competent to give written consent before performing any required steps.

Patient grouping:

All patients will receive perfect professional non-surgical periodontal therapy in form of scaling and root planning and oral hygiene instructions will be given to the patients. Pre-operative periapical x-ray on the area of interest to confirm the integrity of the interproximal bone.The participants were randomly assigned by the toss of a coin into four treatment groups.

Group I It will Include 20 patients and they will be treated with the [LCT] and SCTG. Group II It will Include 20 patients and they will be treated with the [LCT] and MUCODERM.

Group III It will Include 20 patients and they will be treated with the MCAT and SCTG. Group IV It will Include 20 patients and they will be treated with the MCAT and MUCODERM.

Surgical procedure Surgical sites were accurately assessed for each patient. An aseptic field was required for all surgical procedures using povidine iodine. Local anesthesia using 4% articane with 1:100.000 epinephrine was applied for buccal infiltration injection of 1.5 ml and palatal infiltration injection of 0.3 ml. Inferior alveolar nerve block and Lingual nerve block were used for mandibular posterior segment.

Group I-Ⅱ: laterally closed tunnel technique [LCT]

Using a microblade [swan Morton] an internal beveled intrasulcular incisions will be made at the circumferential gingival margin of the affected tooth.

Then specially designed tunneling instruments [devmed] will be used through the sulcular incision to create a pouch. The pouch will be extended apically beyond the mucogingival line and extended mesially and distally from the recession defect undermining all the submucosal tissues.

All fibers should be removed in all directions to ensure optimal tissue mobility without tension.

A microsurgical blade will be used at the inner surface of the pouch till sufficient tissue release will be achieved.

Tissue forceps will be used to approximate the mesial and distal margin of the gingiva at the pouch margin.

Perfect root planning will be performed at the denuded root surface to remove the necrotic cementum.

Subsequently, palatal anesthesia will be given to harvest palatal SCTG using deepithelialized free gingival graft (FGG) technique to get a 1 to 1.5 mm thick connective tissue graft.

After harvesting the graft, it will be placed at the prepared pouch after root surface biomodification using EDTA gel 24% for 2 minutes and copious rinsing with saline solution.

SCTG will be pulled using single or mattress sutures and the graft will be fixed mesial and distal at the inner part of the pouch using resorbable suture material [Vicryl suture], then the graft will be sutured around the neck of the CEJ by sling suture 6/0 polypropylene.

Finally, the margin of the pouch will be adapted close to each other over the graft and sutured together using simple interrupted suturing to get complete or partial coverage of the grafted root surface.

In patients with MUCODERM, after the pouch preparation the collagen matrix will be trimmed to a size suitable for the recession defect then it will be soaked in sterile saline solution for 5 to 10 minutes to allow collagen expansion.

After saturation, the MUCODERM will be inserted into the pouch and sutured in the same way as SCTG.

Patients will be instructed not to brush the surgical site for 14 days and will be ensured to use 0.1% chlorhexidine mouth rinse twice daily for 1 minute each, they will resume brushing after 14 days from the surgery.

Palatal sutures will be removed after 7 days from the surgery, while the sutures at the surgical site will be removed between 14 to 21 days post-surgery. At that time the patients will be instructed to use an ultra-soft toothbrush at the surgical site. Recall professional teeth cleaning will be scheduled 1, 3, 6 months postoperatively.

Group Ⅲ-Ⅳ Modified coronally advanced tunnel technique [MCAT]

The MCAT will be used to treat a single isolated recession defect as the following:

A microsurgical blade [swan Morton] will be used to perform supraperiosteal sulcular incisions at the buccal gingiva of the affected tooth.

Supraperiosteal incisions will be extended to the mucosal level beyond the MGJ to allow sufficient tissue mobility and release.

A Specially designed tunneling knifes with special angles will be used to avoid flap perforation.

The tunnel will be extended in all directions around the recession defect to create a sufficient pouch for connective tissue graft stabilization.

The interdental papilla tunneling adjacent to the defect will be a critical step for technique success. Full thickness tunnel preparation at the papillary region will be done and the papilla will be completely detached from the underlying periosteal layer using mini elevator to avoid tearing.

Then perfect root planning will be performed at the denuded root surface to remove the necrotic cementum at the accessible recession defect.

Subsequently palatal anesthesia will be given to harvest palatal SCTG using deepitheliailized free gingival graft (FGG) technique to get 1 to 1.5 mm thick connective tissue graft.

After harvesting the graft, it will be placed at the prepared pouch after root surface biomodification using EDTA gel 24% for 2 minutes and copious rinsing with saline solution.

SCTG will be pulled using single or mattress sutures and the graft will be fixed mesial and distal at the inner part of the pouch using resorbable suture material [Vicryl suture], then the graft will be sutured around the neck of the CEJ by sling suture 6/0 polypropylene.

After SCTG adaptation, the entire gingival complex will be moved in coronal direction using vertical mattress suture anchored apically at the palatal gingiva.

In patients with porcine-derived collagen matrix( MUCODERM), after the pouch preparation, the collagen matrix will be trimmed to size suitable for the recession defect then it will be soaked in sterile saline solution for 5 to 10 minute to allow collagen expansion.

After saturation the MUCODERM will be inserted into the pouch and sutured in the same wayas SCTG.

Patients will be instructed not to brush the surgical site for 14 days and will be ensured to use 0.1% chlorhexidine mouth rinse twice daily for 1 minute each, they will resume brushing after 14 days from the surgery.

Palatal sutures will be removed after 7 days from the surgery, while the sutures at the surgical site will be removed between 14 to 21 days post-surgery. At that time the patients will be instructed to use ultra-soft toothbrush at the surgical site. Recall professional teeth cleaning will be scheduled 1, 3, 6 months post operatively.

Clinical assessment The following parameters will be measured at the start of the study as well as 3 months and 6 months after the surgery.

Recession depth RD Pink esthetic score PES Root coverage esthetic score RES The mean Root Coverage %RC Gingival Index GI Clinical attachment level CAL Pocket depth PD Keratinized tissue width KTW

ELIGIBILITY:
Inclusion Criteria:

* No systemic diseases or Pregnancy.
* Smoking < 10 cigarettes/day.
* Full mouth plaque score <15%.
* Full mouth bleeding score <15%.
* Presence of isolated gingival recession defect >2 mm in depth
* No interproximal attachment loss.
* No history of previous mucogingival surgeries.

Exclusion Criteria:

* Sever interproximal alveolar bone loss.
* Pregnancy and lactation.
* Heavy smokers.
* Uncontrolled diabetic patients.
* Immunocompromised patients.
* Prosthetic crown at the experimental site.
* Teeth with cervical caries or abrasion.
* Presence of infection or gingival abscess related to the surgical area.
* Bad oral hygiene.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Gingival Recession Depth (RD) | 6 months
  measured as the distance from the CEJ to the gingival margin.

SECONDARY OUTCOMES:
Complete Root Coverage (CRC) | 6 months
  At 6 months follow up the complete root coverage for control and test group were calculated in % , each group.
Mean Root Coverage (MRC) | 6 months
  The mean root coverage % achieved in control group and test group at baseline, 3 months and 6 months with each group.
Gingival Biotype Thickness | 6 months
  Measured 3mm apically from the free gingival margin at the mid buccal aspect of the tooth.
Apico-coronal Width of Keratinized Tissue (KTW) | 6 months
  measured as the distance from the mucogingival junction to the gingival margin, with the mucogingival junction location determined using a visual method with Schiller's Potassium Iodide Solution
Root coverage Esthetic Score (RES) | 6 months
  The RES system evaluated five variables 6 months following surgery: GM, marginal tissue contour (MTC), soft tissue texture (STT), MGJ alignment,and gingival color (GC)
  GM.Zero points=failure of root coverage (gingival margin apical or equal to the baseline recession); 3points=partial root coverage; 6 points=CRC MTC.Zero points=irregular gingival margin (doesnot follow the CEJ); 1 point=proper marginal contour/scalloped gingival margin (follows the CEJ).
  STT.Zero points=scar formation and/or keloid-like appearance; 1 point=absence of scar or keloid formation MGJ.Zero points=MGJ not aligned with the MGJ of adjacent teeth; 1 point=MGJ aligned with the MGJ of adjacent teeth.
  GC.Zero points=color of tissue varies from gingival color at adjacent teeth; 1 point=normal color and integration with the adjacent soft tissues.
  The ideal esthetic score was 10
Pocket Probing Depth | 6 months
  Measured as the distance from the gingival margin to the base of gingival sulcus
Clinical Attachment Level | 6 months
  Measured as Gingival Recession Depth+Probing Depth
Plaque Index (PI) | 6 months
  Silness and Loe 1964
  PI=0 score given when the gingival area of the tooth surface is literally free of plaque.
  PI=1 represents the situation where the gingival area is covered with a thin film of plaque which is not visible,but which is made visible PI=2 score given when the deposit is visible PI=3 is reserved for the heavy (1-2mm.thick) accumulation of soft matter.
Gingival Index (GI) | 6 months
  Loe and Silness 1963
  The criteria are: 0= Normal gingiva; 1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.
  A score from 0.1-1.0 = mild inflammation; 1.1-2.0 = moderate inflammation from, and 2.1-3.0 signifies severe inflammation
Bleeding Index (BI) | 6 months
  Ainamo and Bay 1975 It is performed through gentle probing of the orifice of the gingival crevice. If bleeding occurs within 10 seconds a positive finding is recorded and the number of positive sites is recorded and then expressed as a percentage of the number of sites examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Elmansura, Egypt

REFERENCES:
- [Derived] ElBana A, Saleh W, Youssef J. Comparative evaluation of the laterally closed tunnel technique with connective tissue graft and collagen matrix for treating localized type 1 gingival recession: a randomized, controlled clinical trial. BMC Oral Health. 2026 Jan 6;26(1):184. doi: 10.1186/s12903-025-07515-9. PMID 41495722
- [Derived] Elbana A, Saleh W, Youssef J. Comparing Connective Tissue Grafts and Collagen Matrix in Modified Coronally Advanced Tunnel Technique for RT1 Gingival Recession: A Randomized Controlled Clinical Trial. BMC Oral Health. 2025 Jun 3;25(1):893. doi: 10.1186/s12903-025-06259-w. PMID 40462003